CLINICAL TRIAL: NCT00005713
Title: Improving Care for Minority Children With Asthma: Professional Education in Public Health Clinics
Brief Title: Childhood Asthma Program in NYC Health Department Clinics
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CUMC ID unknown (4922); R01HL045304 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Continuing, preventative care for asthma: Low-income children with asthma will receive continuing, preventive care for asthma with trained staff in New York City Bureau of Child Health clinics
  Interventions: Behavioral: Continuing, preventative care

INTERVENTIONS:
Behavioral: Continuing, preventative care — Training for intervention clinic staff was based on National Asthma Education and Prevention Program guidelines for the diagnosis and management of asthma, and included screening to identify new cases and health education to improve family management.

SUMMARY:
To demonstrate that the New York City Department of Health Child Health Clinics could improve the health status of Black and Hispanic children with asthma by providing them with a comprehensive system of continuity of care that included pharmacologic treatment, family health education and community outreach.

Recent studies have shown that lack of continuing primary care for asthma is associated with increased levels of morbidity in low-income minority children. Although effective preventive therapy is available, many African-American and Latino children receive episodic treatment for asthma that does not follow current guidelines for care. To see if access, continuity, and quality of care could be improved in pediatric clinics serving low-income children in New York City, we trained staff in New York City Bureau of Child Health clinics to provide continuing, preventive care for asthma.

DETAILED DESCRIPTION:
BACKGROUND:

The study was part of a demonstration and education initiative "Interventions for Control of Asthma Among Black and Hispanic Children" which was released by the NHLBI in June 1989.

DESIGN NARRATIVE:

To develop this comprehensive care system, the investigators provided training for Health Department physicians and nurses in up-to-date methods of diagnosing asthma, and providing clinical care and health education to patients and families as part of a series of regular 20 minute patient visits. Nurses and public health assistants were also trained to supplement this by teaching the Open Airways self-management program to groups of families. A 24-hour telephone advice service for families of asthma patients was staffed by trained Health Department physicians.

The intervention was based on social cognitive theory, especially self-regulation. In Phase I, the Health Department medical and nursing staffs were taught by Columbia University faculty with reinforcement by Health Department physician and nurse supervisors. Self-regulation was fostered in physicians by use of an Asthma Visit Record and in families by use of an Asthma Diary. Seven pairs of matched clinics were randomized to be controls or receive the intervention. The following hypotheses were tested: that a comprehensive system of continuity of care, including medical care, family health education and community outreach would (1) increase staff confidence to diagnose and treat childhood asthma; (2) attract and retain families who had children with asthma in continuing care relationships in the Health Department clinics; and (3) improve the health status of patients and the quality of life of their families. Phase II tested whether this comprehensive system could be made self-sustaining within the Health Department by having physician and nurse super-visors who took part in Phase I teach the program to staff from a second set of matched clinics. This program had the potential to reach more than 5000 minority children with asthma. If successful it could be generalized to other health departments in the country.

ELIGIBILITY:
Inclusion Criteria

1. Diagnosed with asthma
2. Attending pediatric clinics serving low-income children in New York City

Exclusion Criteria

1. Unable to return to clinics for follow up and treatment

Ages: 1 Month to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with asthma in New York City
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 1990-08; Primary Completion 1997-02 (Actual); Study Completion 1997-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Evans, MD, Principal Investigator — Professor of Emeritus of Clinical Sociomedical Sciences In Pedi, Dept of Sociomedical Sciences
Locations (1):
- Columbia University, New York, New York, United States

REFERENCES:
- [Background] Evans D, Mellins R, Lobach K, Ramos-Bonoan C, Pinkett-Heller M, Wiesemann S, Klein I, Donahue C, Burke D, Levison M, Levin B, Zimmerman B, Clark N. Improving care for minority children with asthma: professional education in public health clinics. Pediatrics. 1997 Feb;99(2):157-64. doi: 10.1542/peds.99.2.157. PMID 9024439